CLINICAL TRIAL: NCT02746367
Title: A Validation Study to Measure the Impact of a Proteomic Assay in Distinguishing Bipolar I Disorder, Bipolar II Disorder, and Major Depressive Disorder in People Presenting With a Major Depressive Episode
Brief Title: Bipolar Proteomic Assay Validation Study
Status: Completed | Type: Observational
Sponsor: Myriad Genetic Laboratories, Inc. (Industry)
Collaborators: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: EP-001
Record Dates: First submitted 2016-04-12; First posted 2016-04-21 (Estimated); Last update posted 2020-05-14 (Actual); Status verified 2019-03

CONDITIONS: Major Depressive Disorder, Bipolar I and Bipolar II
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Telbivudine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood

GROUPS / COHORTS (3):
- MDD: Patients diagnosed with Major Depressive Disorder
  Interventions: Other: Diagnostic test (LDT)
- BPI: Patients diagnosed with bipolar I
  Interventions: Other: Diagnostic test (LDT)
- BPII: Patients diagnosed with bipolar II
  Interventions: Other: Diagnostic test (LDT)

INTERVENTIONS:
Other: Diagnostic test (LDT) — Proteomic assay

SUMMARY:
The purpose of this study is to validate a set of signatures, based on a panel of proteomic markers, that discriminate BDI, BDII, and MDD in people seeking treatment for a depressive episode.

DETAILED DESCRIPTION:
This is a hypothesis-driven confirmatory study to validate the diagnostic signature (model) for distinguishing BDI from MDD that also aims to optimize the models to discriminate BDII from MDD and BDI. A binary classification model, using linear discriminant analysis and based on 13 a priori-defined proteomic markers will aim to distinguish BDI from MDD. An alternative binary classification model based on multiple logistic regression and using 10 a priori -defined proteomic markers will aim for the same result. To improve the predictive performance of the signatures, items from self-report mood rating scales and treatment-emergent changes in proteomic markers will be analyzed. In addition, the study will examine if baseline or early treatment-emergent changes in proteomic markers predict treatment response.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with BDI, BDII, or MDD, confirmed with the Structured Clinical Interview for DSM-5 (SCID).
* Currently depressed for ≥4 weeks and ≤104 weeks, without psychotic features,
* MADRS score ≥ 20 (consistent with at least moderately-severe depression)
* YMRS score ≤ 8 (consistent with the absence of hypomanic symptoms)

Exclusion Criteria:

* At high risk for suicide, defined as a score ≥4 on item 10 of the MADRS
* Current depression has psychotic features, diagnosed with the SCID
* Meeting criteria for severe alcohol, cannabis, or THC use disorders, as defined by DSM-5 and confirmed by the SCID, in the past 3 months, or meeting criteria for other substance use disorders of any severity (eg. cocaine use disorder). For substances other than alcohol, cannabis, and opioids, a positive drug screen at both the screening and baseline visits is also exclusionary. Caffeine and nicotine use disorders of any severity will not be exclusionary.
* Diagnosis of borderline personality disorder, diagnosed with the Zanarini Rating Scale for Borderline Personality Disorder.
* Medical conditions with neurological sequelae (eg. stroke, brain cancer, multiple sclerosis, loss of consciousness > 30 min, HIV)
* Severe chronic pain, at the discretion of the investigator
* Receiving treatment with high-potency immune-modulating medications, such as corticosteroids, chemotherapy, monoclonal antibodies, or disease-modifying agents for arthritis, multiple sclerosis
* Any acute unstable medical illness (at the discretion of the site investigator)
* In MDD patients: strong risk factors for bipolarity, including 1) short (1-3 day) mood elevations not meeting DSM-5 time criteria for hypomania; 2) a family history of BDI or BDII in a first-degree relative; and 3) a history of antidepressant-induced symptoms suggestive of bipolarity, particularly antidepressant-induced hypo/mania.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients seeking treatment for new on-set depression from academic programs and affiliated community mental health facilities (inpatient and outpatient
Sampling Method: Probability Sample
Enrollment: 261 (Estimated)
Dates: Start 2016-03; Primary Completion 2018-11-08 (Actual); Study Completion 2018-11-08 (Actual)

PRIMARY OUTCOMES:
Agreement between the model derived diagnosis (based on panel of serum proteomic markers) and the clinical diagnosis (confirmed by the SCID DSM-5) | Baseline
  Linear discriminant analysis and multiple logistic regression will be used to create three diagnostic models for the proteomic markers (BDI vs MDD, BDI vs BDII and BDII vs MDD). The patient's model diagnosis will be compared to the patient's clinical diagnoses (based on SCID DSM -5) and the proportion of concordant classifications will be calculated.

SECONDARY OUTCOMES:
Self-report clinical rating scales (IDS-SR30, PHQ-9, MDQ, HCL-32 and TEMPS-A) | Baseline, Week 2 and Week 8
  Additional clinical characterization of the patient and their depressive episode will be obtained through analysis of the self-report clinical rating scales and used to optimize the predictive performance of the proteomic signatures.
Changes in proteomic markers at Week 2 and Week 8 | Week 2 and Week 8
  Proteomic markers will be analyzed at weeks 2 and 8 to observe for any treatment-emergent changes to increase the predictive validity of the proteomic signatures.

OTHER OUTCOMES:
Treatment response (> 50% improvement in MADRS score) | Baseline, Week 8
  Distinguish responders from non-responders by measuring MADRS and determine if baseline or treatment-emergent changes in proteomic markers predict treatment response.
Remission (MADRS score < 8) | Baseline, Week 8
  Distinguish remitters from non-remitters by measuring MADRS and determine if baseline or treatment-emergent changes in proteomic markers predict treatment response.
Antidepressant-induced hypo/mania (YMRS score > 12) | Baseline, Week 2, Week 4, Week 6
  Compare incidence of antidepressant-induced hypo/manic episodes (defined as YMRS score > 12) to changes in proteomic markers to predict treatment response.

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - University of Iowa Health Care, Department of Psychiatry, Iowa City, Iowa
  - University of Minnesota (UMN) Department of Psychiatry, Minneapolis, Minnesota
  - Lindner Center of HOPE/University of Cincinnati College of Medicine, Mason, Ohio
  - University of Pittsburgh Western Psychiatric Institute and Clinic, Pittsburgh, Pennsylvania
  - University of Texas Health Science Center, San Antonio, Texas